CLINICAL TRIAL: NCT05918523
Title: A Long-Term Follow-up Study of Participants Exposed to Renal Autologous Cell Therapy From Studies RMCL-002, REGEN-003, REGEN-004
Brief Title: A Long-Term Follow-Up Study of Participants Exposed to REACT
Status: Recruiting | Type: Observational
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Other Study IDs: REGEN-008S1
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Kidney Disease; Chronic Kidney Diseases
Keywords: REACT; DKD; CKD
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research samples (serum/plasma and/or urine) will be collected, frozen, and stored for the future research. Participating participants can opt out of long-term storage of their unused specimens during the informed consent process or at any time during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD patients previously treated with REACT: Participants Exposed to Renal Autologous Cell Therapy from studies RMCL-002, REGEN-003, REGEN-004 (REGEN-008S1).
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — No interventions in this trial

SUMMARY:
The purpose of this study is to evaluate the long-term safety of up to two gelatin-hydrogel formulation REACT injections given 3 to 6 months apart and delivered percutaneously into same kidney on renal function in participants with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
This observational extension study is a multi-center, prospective, non-therapeutic study, where up to 80 participants who have been enrolled and dosed with Renal Autologous Cell Therapy in previous interventional clinical studies (RMCL-002, REGEN-003, REGEN-004) will be monitored for up to five years with alternating in clinic and phone visits.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have received gelatin-hydrogel formulation REACT in a previous trial (RMCL-002, REGEN-003, REGEN-004) for the treatment of chronic kidney disease and completed an end of study visit in their parent trial per protocol.

Exclusion Criteria:

* The participant did not receive REACT in a previous trial for the treatment of chronic kidney disease.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with CKD
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Long-term safety of REACT | 60 months from completion of parent protocol EOS Visit
  Evaluation of the long-term safety of REACT will be assessed via:
  1. Incidence of delayed serious adverse events (SAEs) obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  2. Incidence of delayed biopsy-related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  3. Incidence of delayed injection procedure related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  4. Incidence of delayed investigational product related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.

SECONDARY OUTCOMES:
First Secondary Endpoint: Time from first injection to eGFR <15 mL/min/1.73m² | 60 months from completion of parent protocol EOS Visit
  Time from first injection to eGFR <15 mL/min/1.73m² using the 2009 CKD-EPI serum creatinine equation.
Second Secondary Endpoint: Time from first injection to chronic dialysis. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to chronic dialysis.
Third Secondary Endpoint: Time from first injection to renal transplant. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to renal transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (1):
- Boise Kidney & Hypertension Institute, Meridian, Idaho, United States